CLINICAL TRIAL: NCT01478750
Title: Oro-gastro-intestinal Digestion of Emulsified Fat and How This Digestion Relates to Colloidal Stability and Physiological Responses
Brief Title: Oro-gastro-intestinal Digestion of Emulsified Fat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Top Institute Food and Nutrition (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NL27994.068.09
Record Dates: First submitted 2011-11-14; First posted 2011-11-23 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Obesity
Keywords: obesity; fat; appetite; digestion
MeSH Terms: conditions — Obesity; Platelet Glycoprotein IV Deficiency | interventions — Sunflower Oil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- emulsified fat, orally (Experimental): At 09:00, subjects will ingest the test load, consisting of 460 water and 40 ml sunflower oil, well emulsified with Tween-80
  Interventions: Dietary Supplement: administration of fat (sunflower oil), emulsified; Procedure: Insertion of nasoduodenal tube
- intragastric administration of fat (Experimental): At 09:00, subjects will receive the load, consisting of 460 water and 40 ml sunflower oil, well emulsified with Tween-80 intragastrically
  Interventions: Dietary Supplement: administration of fat (sunflower oil), emulsified; Procedure: Insertion of nasoduodenal tube
- intraduodenal administration of fat (Experimental): At 09:00, subjects will receive the load, consisting of 460 water and 40 ml sunflower oil, well emulsified with Tween-80 intraduodenally
  Interventions: Dietary Supplement: administration of fat (sunflower oil), emulsified; Procedure: Insertion of nasoduodenal tube
- intragastric, non-emulsified fat (Experimental): At 09:00, subjects will receive the load, consisting of 460 water and 40 ml sunflower oil, non emulsified, intragastrically
  Interventions: Dietary Supplement: administration of fat (sunflower oil), emulsified; Procedure: Insertion of nasoduodenal tube

INTERVENTIONS:
Dietary Supplement: administration of fat (sunflower oil), emulsified — 40 ml sunflower oil, in the presence of the emulsifier tween-80.
Procedure: Insertion of nasoduodenal tube — A nasoduodenal tube is inserted to enable collection of gastric and duodenal aspirates of 2 mL each, to determine gastrointestinal digestion of fat
  Other Names: nasoduodenal intubation; nasoduodenal catheter

SUMMARY:
Interaction of fat with the mouth, stomach and intestine will trigger physiological responses that will impact on the digestion, gut transit time and absorption of fat. These responses will also influence and contribute to regulation of food intake and satiety. No systematic research on understanding how the physiological-chemical properties of food affect the digestion and absorption of lipids has been carried out previously. Studies have shown that the release of free fatty acids triggers the fat-related responses. The investigators hypothesize that the release of fatty acids depends on the colloidal state of the fat, which changes progressively due to the pH changes and enzyme activities in the mouth, stomach and intestine.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form
2. Sex: male or female
3. Age: 18-55 years
4. Body Mass Index (BMI): 18-29 kg/m2
5. Based on medical history and previous examination, no gastrointestinal complaints can be defined.

Exclusion Criteria:

1. Evidence of severe cardiovascular, respiratory, urogenital, gastrointestinal/ hepatic, hematological/immunologic, HEENT (head, ears, eyes, nose, throat), dermatological/-connective tissue, musculoskeletal, metabolic/nutritional, endocrine, neurological/-psychiatric diseases, allergy, major surgery and/or laboratory assessments which might limit participation in or completion of the study protocol
2. Gastrointestinal or hepatic disorders influencing gastrointestinal absorption or transit
3. Use of psychotropic drugs, including: benzodiazepines. Concomitant medication that can increase gastric pH (e.g. antacids, proton pump inhibitors, prostaglandins, anticholinergic agents, H2-receptor antagonists), or alter gastric emptying (e.g. metoclopramide, cisapride, domperidone and erythromycin, anticholinergics, tricyclic antidepressants, narcotic analgetics, adrenergic agents, calcium channel blockers), or alter intestinal transit (e.g., loperamide, chemical/osmotic/bulk laxatives) or influence satiety/energy intake (e.g. sibutramine, glucocorticoids, anabolic steroids), except oral contraceptives
4. Pregnancy, lactation, wish to become pregnant during study, or having a positive pregnancy test at inclusion
5. Reported unexplained weight loss/gain of more than 2 kg in the month before the study enrollment
6. Score > 9 on Factor 1 (dietary restrained) of the Dutch translation of the Three Factor eating Questionnaire (TFEQ) [17]
7. Blood donations less than three months previous to study enrollment, and for three months following participation
8. One or more of the following dietary habits: medically prescribed diets, weight reduction diets, or vegetarian/macrobiotic/biologically dynamic food habits. Administration of investigational drugs in the 180 days prior to the study
9. Major abdominal surgery interfering with gastrointestinal function (uncomplicated appendectomy, cholecystectomy and hysterectomy allowed, and other surgery upon judgement of the principle investigator)
10. Premenstrual syndrome, dieting (medically prescribed, vegetarian, diabetic, biological dynamic)
11. Excessive alcohol consumption (>20 alcoholic consumptions per week)
12. Smoking
13. Self-admitted HIV-positive state

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2009-12; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Appearance of free fatty acids in the duodenum | In the first 180 min after administration of test product
  The appearance of free fatty acids in the duodenum will be assessed during the 180 min following ingestion of the test product.

SECONDARY OUTCOMES:
Colloidal stability of fat | In the first 180 min after administration of test product
  Droplet size, flocculation, aggregation, coalescence) in samples from the oral, gastric and duodenal compartment will be determined during the 180 min following ingestion of the test product.

CONTACTS AND LOCATIONS:
Overall Officials: Freddy Troost, PhD, Principal Investigator — Maastricht University Medical Centre
Locations (1):
- Maastricht University Medical Centre, Maastricht, Netherlands